CLINICAL TRIAL: NCT04882774
Title: Telemonitoring to Treat Group 2 Pulmonary Hypertension: A Personalized Approach
Brief Title: Telemonitoring to Treat Group 2 Pulmonary Hypertension
Acronym: RECAPTURE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: never opened to enrollment because it was never funded
Sponsor: Mardi Gomberg -Maitland MD, MSc (Other)
Collaborators: Ohio State University (Other); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Sponsor-Investigator, Mardi Gomberg -Maitland MD, MSc, Director, Pulmonary Hypertension Program, George Washington University
Organization: George Washington University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RECAP001
Record Dates: First submitted 2021-04-27; First posted 2021-05-12 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Hypertension Due to Left Heart Disease
MeSH Terms: interventions — treprostinil

STUDY DESIGN:
Intervention Model Description: 32 week study in 30 subjects. Those who meet certain hemodynamic criteria at Week 16 will begin study drug and continue diuresis protocol while the remaining participants continue with the diuresis protocol only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fluid Management (No Intervention): Fluid management protocol only
- Oral Treprostinil (Experimental): Drug - oral treprostinil
  Interventions: Drug: Treprostinil Diolamine

INTERVENTIONS:
Drug: Treprostinil Diolamine — Oral treprostinil 0.125 mg TID titrated as clinically indicated and tolerated to a maximum of 6 mg TID
  Arms: Oral Treprostinil

SUMMARY:
This study aims to decrease elevated pressure in the lungs of patients with pulmonary hypertension from left heart with elevated pulmonary vascular resistance by utilizing aggressive fluid management with ReDS Pro System and CardioMEMS device. Participants with persistently elevated pulmonary pressure at Week 16 will begin oral treprostinil in combination with the fluid management plan while those with improved pressures maintain their fluid management plan for an additional 16 weeks.

DETAILED DESCRIPTION:
This study hypothesizes that monitoring with ReDS-Pro System (ReDS), aggressive fluid management, and the CardioMEMS device (a 3-prong approach) will improve CpcPH (combined pre and post capillary pulmonary hypertension) hemodynamics (Total Pulmonary Resistance [TPR] and mPAP). For patients who continue to have an elevate pulmonary vascular resistance (TPR) at Week 16, with ReDS, aggressive fluid management, and the CardioMEMS device should allow successful titration of oral treprostinil by preventing titration related pulmonary edema and by improving hemodynamics, activity monitoring and six minute walk test (6MWT) after 16 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily gives informed consent to participate in the study.
* The subject is 18 to 85 years of age (inclusive) at Baseline (i.e., date of providing written informed consent).
* The subject has a diagnosis of heart failure with a LVEF ≥45% by ECHO completed prior to randomization.
* The subject has a CardioMEMS device implanted as standard of care for a minimum of 30 days at Baseline.
* The subject has pulmonary function tests conducted within 12 months of Baseline or to confirm the following:

  1. Total lung capacity is ≥ 60% of the predicted value.
  2. Forced expiratory volume at 1 second (FEV1) is ≥50% of the predicted value.
  3. Diffusing capacity of the lungs for carbon monoxide (DLCO) is ≥ 32% of the predicted value (unadjusted or adjusted for alveolar volume).
* Subjects should be on maximally tolerated HFpEF therapies (e.g., ACE inhibitors, ARBs, beta blockers, SLG2 inhibitors) for ≥30 days prior to enrollment unless contraindicated. The exception is with changes of anticoagulants and/or diuretics; these medications should not be newly started or stopped within 14 days of enrollment and no healthcare provider prescribed dose change should occur within 7 days of enrollment, with the exception of the withholding of doses of anticoagulants for the conduct of the RHC when required.
* In the opinion of the Investigator, the subject is able to communicate effectively with study personnel, and is considered reliable, willing, and likely to be cooperative with protocol requirements, including attending all study visits.
* Subjects on chronic medications (e.g. inhaled corticosteroids, long-acting beta2-adrenergic agonist, long-acting muscarinic antagonists, combination inhaled drugs, anti-inflammatory drugs, oral/parenteral corticosteroids, or biologic agents) for any underlying respiratory condition must be on a stable dose for ≥30 days prior to randomization.

Exclusion Criteria:

* The subject is pregnant or lactating.
* In the opinion of the Principal Investigator, the subject has a primary diagnosis of PH other than WHO Group 2 PH.
* The subject has shown intolerance or significant lack of efficacy to a prostacyclin or prostacyclin analogue that resulted in discontinuation of therapy or inability to effectively titrate that therapy.
* The subject has received PAH therapies, including prostacyclin therapy (i.e., epoprostenol, treprostinil, iloprost, or beraprost; except for acute vasoreactivity testing), nonprostanoid IP receptor agonist (selexipag), ERA, or soluble guanylate cyclase stimulator, within 30 days of enrollment. If the Investigator does not intend to keep a subject on their PDE5-I therapy, it must be stopped at least 30 days prior to enrollment. Intermittent use of a PDE5-I (≤3 times per week) to treat erectile dysfunction is permitted.
* The subject has been hospitalized for a cardiopulmonary indication within 30 days of randomization.
* The subject had a myocardial infarction within 90 days of enrollment.
* The subject had cardiac resynchronization therapy within 90 days of enrollment or anticipated resynchronization therapy during the study treatment period.
* The subject has liver function tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) greater than 3 times the upper limit of normal at Screening, clinically significant liver disease/dysfunction per Investigator's clinical judgement, known Child-Pugh Class C hepatic disease or noncirrhotic portal hypertension.
* The subject has uncontrolled systemic hypertension, defined as a systolic blood pressure >160 mmHg or a diastolic blood pressure >110 mmHg at Baseline on more than one occasion during screening.
* The subject has a systolic blood pressure <100 mmHg at Baseline.
* The subject has a resting heart rate >110 beats per minute at Baseline.
* The subject has sarcoidosis or cardiac amyloidosis.
* The subject has a known history of any LVEF less than 40% by ECHO within 3 years of enrollment. Note: a transient decline in LVEF below 40% that occurred and recovered more than 6 months before the start of Screening and was associated with an acute intercurrent condition (e.g., atrial fibrillation) is allowed.
* The subject has hemodynamically significant valvular heart disease as determined by the Investigator, including:

  1. Greater than mild aortic and/or mitral stenosis
  2. Severe mitral and/or aortic regurgitation (>Grade 3)
* The subject has a body mass index >45 kg/m2.
* The subject has any musculoskeletal disorder (e.g., arthritis affecting the lower limbs, recent hip or knee joint replacement, artificial leg), or has any other condition that would likely be the primary limit to ambulation as opposed to the disease under study.
* The subject has end-stage renal disease requiring/receiving dialysis.
* The subject has used any investigational drug/device, or participated in any investigational study, within 30 days prior to the Baseline visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with normal lung impedance as measured by the ReDS vest in Ohms at Week 16 | 16 weeks
  Number of participants reaching normal lung impedance (< 34 Ω) based on ReDS vest management.
Number of participants with normal total pulmonary resistance as measured by CardioMEMS in Woods Units at Week 16 | 16 weeks
  Number of participants reaching normal total pulmonary resistance (< 5 Woods Units) as measured by CardioMEMS.
Number of participants reaching normal lung impedance with oral treprostinil at Week 32 | 16 weeks
  Number of participants reaching normal lung impedance (<34 Ω) from Week 16 to Week 32 with oral treprostinil administration.
Number of participants reaching normal total pulmonary resistance with oral treprostinil at Week 32 | 16 weeks
  Number of participants reaching normal total pulmonary resistance (goal < 5 U) from Week 16 to Week 32 with oral treprostinil administration.
Number of participants decreasing six-minute walk distance with oral treprostinil at Week 32 | 16 weeks
  Number of participants with a six-minute walk distance decrease of >15% from Week 16 to Week 32 with oral treprostinil administration.
Number of participants maintaining normal lung impedance as measured by the ReDS vest at Week 32 | 16 weeks
  Number of participants maintaining normal lung impedance (< 34 Ω) from Week 16 to Week 32 as measured by ReDS vest.
Number of participants maintaining total pulmonary resistance as measured by CardioMEMS at Week 32 | 16 weeks
  Number of participants maintaining normal TPR (< 5 U) from Week 16 to Week 32 as measured by CardioMEMS.

SECONDARY OUTCOMES:
WHO Functional Class | 32 weeks
  Change in Functional Class (FC) Week 16, 32.
Change in cardiac output | 32 weeks
  Change in cardiac output (L/min) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in cardiac index | 32 weeks
  Change in cardiac index (L/min/m2) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in right ventricular stroke volume | 32 weeks
  Change in right ventricular stroke volume (mL) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in stroke volume index | 32 weeks
  Change in stroke volume index (mL/m2) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in elastance | 32 weeks
  Change in elastance (mmHg/mL) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in compliance | 32 weeks
  Change in compliance (mL/mmHg) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in right ventricular power | 32 weeks
  Change in right ventricular power (W) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in cardiac efficiency | 32 weeks
  Change in cardiac efficiency (mL/mmHg) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in right ventricular stroke work | 32 weeks
  Change in right ventricular stroke work (mmHg/mL) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in stroke work index | 32 weeks
  Change in stroke work index (g x m/m2) as measured by CardioMEMS from Baseline to Week 16, 32.
Change in NT-proBNP | 32 weeks
  Change in N-terminal pro-brain natriuretic peptide (NT-proBNP) levels from Baseline to Week 16, 32.
Kansas City Cardiomyopathy Questionnaire | 32 weeks
  Improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) at Baseline to Week 16 and baseline to Week 32. Scores are scaled from 0 to 100 and summarized in quartiles representing health status with higher scores indicating better status: 0 to 24=very poor to poor; 25 to 49=poor to fair; 50 to 74=fair to good; and 75 to 100= good to excellent.
Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire | 32 weeks
  Improvement in PAH-SYMPACT at Baseline to Week 16, Baseline to Week 32. Measured using the Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire with higher scores indicating greater symptom severity or worse impact: scale of 0=no, 1=mild, 2=moderate, 3=severe, and 4=very severe.
Number of participants with heart failure exacerbation | 32 weeks
  Adjudicated hospitalization or emergency department visits due to a heart failure decompensation.
Six-minute walk test | 32 weeks
  Decrease in 6MWT >15% from Baseline (or too ill to walk) directly related to disease under study at 2 consecutive visits on different days.
Number of participants who experienced mortality | 32 weeks
  Heart failure related deaths and all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Mardi Gomberg-Maitland, MD, Principal Investigator — George Washington University; Raymond Benza, MD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - George Washington University, Washington D.C., District of Columbia
  - Ohio State University, Columbus, Ohio
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No